CLINICAL TRIAL: NCT05438719
Title: An Interventional, Multi-center Investigation of the MOTUS Total Joint Replacement
Brief Title: MOTUS Total Joint Replacement Investigational Device Exemption Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 3Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOTUS IDE
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Spine Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MOTUS (Experimental): All subjects will be treated with the MOTUS Total Joint Replacement
  Interventions: Device: MOTUS Total Joint Replacement

INTERVENTIONS:
Device: MOTUS Total Joint Replacement — The MOTUS Total Joint Replacement is indicated for the biomechanical reconstruction and stabilization of a spinal motion segment following decompression at one lumbar level from L1/L2 to L5/S1 for skeletally mature patients due to symptomatic lumbar degeneration with or without foraminal or recess spinal stenosis confirmed by radiographic imaging (CT, MRI, X-rays), with no more than a Grade 1 spondylolisthesis at the involved level.

SUMMARY:
This study is designed to collect safety and efficacy data on patients who plan to undergo a single-level total joint replacement of the lumbar spine using the MOTUS device (MOTUS Total Joint Replacement procedure) to demonstrate noninferiority to lumbar interbody fusion with respect to composite endpoints.

DETAILED DESCRIPTION:
A multi-center (up to 20 investigational sites), prospective, non-blinded investigation of the MOTUS Total Joint Replacement (TJR) device. These data will be compared to a lumbar interbody fusion (transforaminal lumbar interbody fusion [TLIF] or posterior lumbar interbody fusion [PLIF]) control group enrolled in a separate real world evidence (RWE) study. Balance between groups will be achieved through sub classification using propensity scores by a blinded statistician.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 21-80 (inclusive) with at least 3 years of life expectancy
2. The subject has a primary diagnosis of symptomatic lumbar degeneration with or without foraminal or recess stenosis of the lumbar spine at a single level from L1/L2 to L5/S1 confirmed by subject history and radiographic imaging (CT, MRI, X- rays) with no more than a Grade 1 (<25% translation) spondylolisthesis. Symptomatic lumbar degeneration that may be associated with a co-morbid condition such as:

   1. Herniated nucleus pulposus
   2. Scarring/thickening of the ligamentum flavum, annulus fibrosus, or facet joint capsule
   3. Facet joint degeneration/osteophyte formation
   4. Spondylosis (defined by the presence of osteophytes)
   5. Disc degeneration and/or annular degeneration; and/or
   6. Lumbar stenosis defined by spinal cord or nerve root compression
3. Exhausted conservative treatment (e.g. bed rest, physical therapy, medications, TENS (transcutaneous electrical nerve stimulation), manipulation, and/or spinal injections) for at least 3 months or has a neurologic emergency
4. Preoperative Oswestry Disability Index score ≥ 40/100 at baseline
5. Psychosocially, mentally, and physically able and willing to fully comply with this protocol including adhering to follow-up schedule and requirements and filling out forms
6. Signed informed consent.

Exclusion Criteria:

1. More than one vertebral level requiring treatment
2. Previous instrumented surgery (i.e.: anterior disc replacement, spinal fusion, interspinous device, etc.) at the index lumbar level or an adjacent level
3. Degenerative or lytic spondylolisthesis greater than Grade 1 (25% translation)
4. Rotatory scoliosis at the index level
5. Congenital bony and/or spinal cord abnormalities at the index level
6. Subcaudal defect, disrupting the integrity of the pedicle
7. Clinically compromised vertebral bodies at the index level due to current or past trauma, e.g., by the radiographic appearance of the fracture callus, malunion or nonunion
8. Disrupted anterior longitudinal ligament at the index level
9. Overlying thoracolumbar kyphosis (greater than or equal to 15 degrees) within one level (includes target and adjacent level) of the level to be treated
10. Back pain of unknown etiology without leg pain
11. Severe spondylosis at the level to be treated as characterized by any of the following:

    1. Autofusion (solid arthrodesis) determined radiographically (CT)
    2. Totally collapsed disc, or
    3. Vertebral body that cannot be mobilized
12. Known allergy to cobalt, chromium, molybdenum, nickel, polyethylene, titanium, or vitamin E
13. Unable to undergo an MRI scan, CT scan or other radiograph assessments
14. Osteopenia: The SCORE/MORES will be utilized for all females age <50 and males age <55 to screen if a DEXA scan is indicated. If SCORE/MORES value ≥ 6, then a DEXA scan is required. A DEXA scan is indicated for all females age ≥50 and all males age ≥55. If DEXA is required, exclusion will be defined as a DEXA bone density measured T score ≤ -1. An existing DEXA is allowed if completed within 6 months of subject screening;
15. Has history of any endocrine or metabolic disorder known to affect osteogenesis (e.g.: Paget's disease, renal osteodystrophy, Ehler-Danlos syndrome, or osteogenesis imperfecta)
16. Insulin-dependent diabetes mellitus
17. Lactating, pregnant or interested in becoming pregnant in the next 3 years
18. Active infection - systemic or local
19. Any medical condition requiring treatment with any drug known to potentially interfere with bone/soft tissue healing or receiving radiation therapy that is expected to continue for the duration of the study
20. Body Mass Index > 40
21. Recurrent history of deep vein thrombosis, symptoms of arterial insufficiency, or thromboembolic disease
22. Systemic disease including Lupus disease, Reiter's disease, Rheumatoid disease, AIDS, HIV, hepatitis or autoimmune disease that requires immunosuppressive therapy, including biologics, for systemic inflammation
23. Spinal tumor
24. Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
25. Any degenerative muscular or neurological condition that would interfere with evaluation of outcomes, including but not limited to Parkinson's disease, amyotrophic lateral sclerosis (ALS), or multiple sclerosis
26. Has chronic or acute renal and/or hepatic impairment and/or failure or prior history of renal and/or hepatic parenchymal disease
27. Has a Waddell Signs of Inorganic Behavior score of 3 or greater
28. In the opinion of the investigator, the subject has a behavioral, cognitive, social or medical problem that may interfere with the assessment of the safety or effectiveness of the device
29. Current or recent history of chemical/alcohol abuse or dependency using standard medical definition of DSM-5 (Diagnostic and Statistical Manual) code
30. Currently smoking or using tobacco products, including e-cigarette products (e.g., vaping) (Use within 30 days of surgery date is considered 'current')
31. Currently pursuing or in active spinal litigation for medical negligence, or trauma, or workers compensation
32. Is a prisoner, incarcerated, or has been coerced to participate in the study that could impact the validity of results
33. Is currently participating in an investigational therapy (device and/or pharmaceutical) within 30 days prior to entering the study or such treatment is planned during the 24 months following enrollment into the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-06-13 (Estimated); Study Completion 2029-06-13 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Score | 24 months compared to baseline
  Improvement of at least 15 points in ODI score (out of 100). The ODI is a self-reported questionnaire that contains ten sections concerning intensity of pain, lifting, personal care, walking, sitting, sexual function, standing, social life, sleeping and traveling.
Neurological Status | 24 months compared to baseline
  Absence of deterioration in neurological status compared to baseline examinations. Neurological examination will consist of a motor and sensory examination at each in person study visit conducted per physician standard of care. These data will be adjudicated by the Clinical Events Committee (CEC).
Secondary Surgical Intervention (SSI) | 24 month
  Subject success will be determined with the absence of a secondary surgical intervention including revision, re-operation, removal, or supplemental fixation at the index level.
Serious device-related adverse events (SDAE) | 24 month
  Subject success will be determined with the absence of any serious device-related adverse events (SDAE). These data will be adjudicated by the Clinical Events Committee (CEC).

SECONDARY OUTCOMES:
Visual Analog Score (VAS) - Worst Leg | 24 months
  Improvement in VAS - Worst leg of 20mm at 24 months compared to baseline
VAS - Back | 24 months
  Improvement in VAS - Back pain of 20mm at 24 months compared to baseline
ODI | 24 months
  Improvement in ODI of 15 points at 24 months compared to baseline
ODI | 24 months
  Mean change in ODI over time intervals
VAS | 24 months
  Mean change in leg VAS over time intervals
VAS | 24 months
  Mean change in back VAS over time intervals
Radiographically confirmed subsidence | 24 months
  Absence of radiographically confirmed subsidence >5mm

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) | 24 months
  Improvement in PROMIS scores at 24 months relative to the baseline.
Demographics | 24 months
  The study will examine the patient population through descriptive statistics of the demographic variable - age
Demographics | 24 months
  The study will examine the patient population through descriptive statistics of the demographic variable - Body Mass Index (BMI)
Demographics | 24 months
  The study will examine the patient population through descriptive statistics of the demographic variable - gender
Intra-Operative Variables | 24 months
  The study will examine the patient population through descriptive statistics of the intra-operative variable - surgery time.
Intra-Operative Variables | 24 months
  The study will examine the patient population through descriptive statistics of the intra-operative variable - blood loss
Time to first SSI | 24 months
  Time to first SSI including specific actions (removal, revision, replacement, supplemental fixation) at the index or adjacent level

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Todd H. Lanman, MD Inc., Los Angeles, California
  - Steamboat Orthopaedic & Spine Institute (SOSI), Steamboat Springs, Colorado
  - Spine an Orthopedic Center, Deerfield Beach, Florida
  - Florida Orthopaedic Institute, Temple Terrace, Florida
  - Strenge Spine Institute, Paducah, Kentucky
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Upstate Ortho, East Syracuse, New York
  - NYU Langone, New York, New York
  - Pinehurst Surgical Clinic, Pinehurst, North Carolina
  - Oklahoma Spine Center, Oklahoma City, Oklahoma
  - Center for Sports Medicine and Orthopaedics, Chattanooga, Tennessee
  - Orthopedic San Antonio, San Antonio, Texas
  - The Disc Replacement Center, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Undecided